CLINICAL TRIAL: NCT05407428
Title: An Prospective Study in a Cohort of Amyotrophic Lateral Sclerosis (ALS) Patients Participating in a Phase IIb Drug Study (NCT05357950) to Evaluate the Correlation Between Oculometric Measurements and ALS Functional Rating Scale (ALSFRS-R)
Brief Title: A Prospective Study to Evaluate the Correlation Between Oculometric Measurements and Clinical Endpoints in ALS Patients
Status: Completed | Type: Observational
Sponsor: NeuraLight (Industry)
Responsible Party: Sponsor
Other Study IDs: NL/ALS/2022-2
Record Dates: First submitted 2022-05-29; First posted 2022-06-07 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: NeuraLight software-based platform — NeuraLight is an investigational software-based platform that is used for assessment and evaluation of neurological conditions including ALS patients

SUMMARY:
This is a prospective study in a cohort of about 45 patients with ALS participating in the Neurosense PrimeC drug study (NCT05357950).

This study aims to evaluate the correlation between oculometric measures and clinical endpoints. Subjects will be evaluated every 2 months during a time period of 18 months. The evaluations will include ALSFRS-R examination, as well as an oculometric evaluation for eye movements.

DETAILED DESCRIPTION:
This is an observational prospective study in a cohort of about 45 patients with ALS participating in the Neurosense PrimeC drug study (NCT05357950), which is a Phase IIb, Randomized, Prospective, Double-Blind, Placebo-Controlled Study, to Evaluate Safety, Tolerability and Efficacy of PrimeC in Subjects with ALS. The subjects are males or females with familial or sporadic ALS of no more than 30 months disease duration, who meet the inclusion criteria of the PrimeC drug study, provide a signed an Informed consent and are willing and able to comply with study's procedures including follow-up visits.

This study is designed to evaluate the correlation between oculometric measures and the Revised Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS-R). Subjects will be evaluated every 2 months during a time period of 18 months. The evaluations will include an ALSFRS-R examination by a certified neurologist and other tests. In addition, all patients will undergo a NeuraLight session for oculometric evaluation along with eye-tracking recordings. All assessments will be performed during a clinic visit unless authorized to be conducted remotely.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and willing to sign an informed consent form (ICF)
* Males or females between the ages of 18 and 75 years of age, inclusive
* Diagnosis of familial or sporadic ALS (defined as meeting the laboratory-supported probable, probable, or definite criteria for a diagnosis of ALS according to the Gold Coast criteria)
* Disease duration after first symptom (muscle weakness) less than 30 months prior to screening
* Pre-enrollment ALSFRS-R slope from disease onset ≥ 0.3 points per month
* ALSFRS-R at screening ≥ 25
* Item 3 (swallowing) in ALSFRS-R ≥ 3
* Subjects may be treated in parallel with Riluzole and/or Edaravone and/or Sodium Phenylbutyrate; 30 days of stable use prior to enrollment is required
* Upright slow vital capacity (SVC) ≥ 60% of predicted for age, height, weight and sex at screening according to the GLI-2012
* 18 < BMI < 30
* A caregiver (if one is needed)
* Female subjects must be post-menopausal (≥ 1 year) OR sterilized, OR if of childbearing potential (i.e., females who have had their first period unless they are anatomically or physiologically incapable to become pregnant), must have a negative pregnancy test, and agree to use contraceptive drugs or devices (e.g., diaphragm plus spermicide, or oral contraceptives) for the duration of the study and 10 weeks after the last treatment dose AND require male partners to use a condom during sexual intercourse

Exclusion Criteria:

* A past history of adverse reaction/hypersensitivity to either NSAIDs, celecoxib or fluoroquinolones, ciprofloxacin
* Any known clinically significant abnormal gastric mucosal erosion, ulcer or tumor or/and GI disorder and/or bariatric surgery Known history of clinically significant impairment of renal function (creatinine ≥ 1.5)
* Known or suspected symptomatic congestive heart and/or coronary heart disease, previous history of myocardial infarction, uncontrolled arterial hypertension, or rhythm abnormalities requiring permanent treatment
* Known history of QT/QTc prolongation, Torsade de pointes (TdP) (e.g. heart failure, hypokalemia, family history of Long QT syndrome) and the use of concomitant medications that prolong the QT/QTc interval
* Known or suspected diagnosis or family history of epilepsy in first degree relatives
* Known predisposition to tendinitis
* Tracheostomy or percutaneous gastrostomy use
* Presence at screening of any medically significant cardiac, pulmonary, musculoskeletal, or psychiatric illness that might interfere with the subject's ability to comply with study procedures or that might confound the interpretation of clinical safety data, including, but not limited to:

  1. Mean systolic blood pressure >160 mm Hg and/or mean diastolic blood pressure >100 mm Hg (measurements taken after a few minutes rest) that persist on 3 successive measurements taken at least 2 minutes apart
  2. NYHA Class II or greater congestive heart failure
  3. Chronic obstructive pulmonary disease or asthma requiring daily use of bronchodilator medications
  4. Poorly controlled or brittle diabetes mellitus
  5. Cognitive impairment, related to ALS or otherwise, sufficient to impair subject's ability to understand and/or comply with study procedures and provide informed consent
* Subject who is treated with chronic aspirin or NSAIDs and is at risk if stopped. Clopidogrel is allowed and can replace Aspirin.
* Any contraindication for ciprofloxacin and celecoxib according to the current prescribing information.
* Female who is pregnant or breastfeeding or with intention of becoming pregnant during the course of the study.
* Any impairment or social circumstance that, in the opinion of the Investigator, would render the subject not suitable to participate in the study.
* Subject, or subject's legal guardian(s) is/are unable to understand the nature, scope, and possible consequences of the study.
* Subject is participating in (or plans to participate in) any other investigational drug trial, or plans to be exposed to any other investigational agent, device and/or procedure, from 30 days prior to Screening through study completion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: About 45 ALS patients, ages 18-75 years with familial or sporadic ALS, according to the Gold Coast Criteria, who are recruited and participating in the PrimeC drug study (NCT05357950)
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Correlation between ALSFRS-R score and its parts with NeuraLight oculometric measurements | 18 months
  The correlation between ALSFRS-R score and its parts with NeuraLight oculometric measurements (R-Square>0.5, p<0.05) according to the measured ALS functional rating scale - revised (ALSFRS-R) at every visit
Feasibility of using NeuraLight system to capture oculometric measures in a cohort of ALS patients | 18 months
  Capturing >50 different oculometric measures in >95% of a cohort of 45 patients
Comparison of NeuraLight extracted oculometric measures with a validated eye-tracking system | 18 months
  Relative root mean square error (RMSE) of NeuraLight's extracted oculometric measures compared with retrieved measurements from a validated eye tracking system <0.1

SECONDARY OUTCOMES:
Using the retrieved data of collected NeuraLight oculometric measures for calibration of prediction models of ALSFRS-R clinical endpoint | 18 months
  Optimization of a feature selection model (Fisher's Linear Discriminant Analysis (LDA)) on NeuraLight oculometric measures used for a logistic regression model of ALSFRS-R with a relative root mean square error (RMSE) of <0.1

CONTACTS AND LOCATIONS:
Overall Officials: Vivian Drory, MD, Principal Investigator — Sackler Faculty of Medicine, Tel Aviv University
Locations (1):
- Sourasky medical center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No
There is not plan to share IPD with other researchers

REFERENCES:
- [Background] Kang BH, Kim JI, Lim YM, Kim KK. Abnormal Oculomotor Functions in Amyotrophic Lateral Sclerosis. J Clin Neurol. 2018 Oct;14(4):464-471. doi: 10.3988/jcn.2018.14.4.464. Epub 2018 Jun 27. PMID 30198218
- [Result] Guo X, Liu X, Ye S, Liu X, Yang X, Fan D. Eye Movement Abnormalities in Amyotrophic Lateral Sclerosis. Brain Sci. 2022 Apr 11;12(4):489. doi: 10.3390/brainsci12040489. PMID 35448020